CLINICAL TRIAL: NCT00674362
Title: A Phase IIIB, Multi-center, Double-blind, Placebo-controlled, Parallel Group, 52-week Study to Evaluate the Safety and Efficacy of Certolizumab Pegol, Administered With DMARDs, in Patients With Low to Moderate Disease Activity Rheumatoid Arthritis
Brief Title: Rheumatoid Arthritis (RA) Moderate to Low Disease Activity Study
Acronym: CERTAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C87076; 2007-000828-40 (EudraCT Number)
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2012-01-18 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2011-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Moderate to Low Disease activity; Certolizumab pegol
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Certolizumab pegol 200 mg (CDP870) (Experimental): Two 200 mg subcutaneous injections at Week 0, Week 2, and Week 4 followed by 200 mg injections every 2 weeks until the last drug administration (Week 22)
  Interventions: Biological: Certolizumab pegol
- Placebo (Placebo Comparator): Two 0.9% saline subcutaneous injections at Week 0, Week 2, and Week 4 followed by 0.9% saline injections every 2 weeks until the last drug administration (Week 22)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Certolizumab pegol — Two 200 mg subcutaneous injections at Week 0, Week 2, and Week 4 followed by 200 mg injections every 2 weeks until the last drug administration (Week 22)
  Other Names: CDP870; Cimzia
  Arms: Certolizumab pegol 200 mg (CDP870)
Biological: Placebo — Two 0.9% saline subcutaneous injections at Week 0, Week 2, and Week 4 followed by 0.9% saline injections every 2 weeks until the last drug administration (Week 22)
  Arms: Placebo

SUMMARY:
To assess the clinical efficacy and safety of certolizumab pegol as add-on therapy with stable-dose disease-modifying antirheumatic drugs (DMARDs) for achieving clinical remission in patients with moderate to low disease activity rheumatoid arthritis

DETAILED DESCRIPTION:
Treatment period starts with a 24-week, double blind, placebo-controlled, randomized period followed by an open label phase until week 52.

In the double blind phase eligible patients will be randomized via an Interactive Voice Response System (IVRS) in a 1:1 ratio to receive either certolizumab pegol (400 mg at Weeks 0, 2 and 4, followed by 200 mg every two weeks) or placebo up to and including Week 22. All patients will continue to receive their Disease Modifying AntiRheumatic Drugs (DMARDs) therapy established before study entry until Week 52. At Week 24, patients will not receive any injection but will be evaluated:

* Non-remitters at Week 24 (patients who did not achieve remission at both Week 20 and Week 24) will be discontinued from the study and may be given the opportunity to enter in an open-label follow-up trial, C87080 [NCT00843778], with certolizumab pegol.
* Remitters (i.e. patients who achieved remission as measured by Clinical Disease Activity Index (CDAI) at both Week 20 and Week 24) will stop their randomized treatment (certolizumab pegol or placebo) and be followed up until Week 52. Remitters who flare up (CDAI ≥11 confirmed at two consecutive visits four weeks apart) between Week 24 and Week 52 will be re-treated with the same dosing regimen of certolizumab pegol (3 administrations of 400mg, given every 2 weeks, followed by 200 mg given every other week) up to and including Week 50.

Remitters who flare up between Week 24 and Week 52 and complete 52-week study period will be allowed to enter open label follow up trial at Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established diagnosis of low to moderate adult rheumatoid arthritis, currently on Disease Modifying AntiRheumatic Drugs (DMARDs) therapy for at least six months and not longer than 10 years

Exclusion Criteria:

* All the concomitant diseases or pathological conditions that could interfere and impact the assessment of the study treatment, or with the safety of the patient
* Previous clinical trials and previous biological therapy that could interfere with the results in the present clinical trial
* Patients must not have received any previous biological therapy for rheumatoid arthritis (RA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (31):
- Austria (2):
  - Graz
  - Vienna
- France (5):
  - Nantes
  - Paris
  - Rennes
  - Rouen
  - Tours
- Germany (11):
  - Bad Nauheim
  - Berlin
  - Erlangen
  - Essen
  - Frankfurt
  - Hamburg
  - Heidelberg
  - Herne
  - Ratingen
  - Vogelsang-Gom
  - Würzburg
- Italy (4):
  - Ferrara
  - Padua
  - Pavia
  - Roma
- Poland (9):
  - Bialystok
  - Bydgoszcz
  - Elblag
  - Lublin
  - Poznan
  - Sopot
  - Szczecin
  - Torun
  - Wroclaw

REFERENCES:
- [Derived] Smolen JS, Emery P, Ferraccioli GF, Samborski W, Berenbaum F, Davies OR, Koetse W, Purcaru O, Bennett B, Burkhardt H. Certolizumab pegol in rheumatoid arthritis patients with low to moderate activity: the CERTAIN double-blind, randomised, placebo-controlled trial. Ann Rheum Dis. 2015 May;74(5):843-50. doi: 10.1136/annrheumdis-2013-204632. Epub 2014 Jan 15. PMID 24431394
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started in June 2008 with subjects from Germany, France, Austria, Italy, and Poland. The primary completion date occurred in May 2010, with an anticipated study completion in December 2010.
Period: Double Blind
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Started | 96 | 98
Completed | 84 | 80
Not Completed | 12 | 18
Not completed — Adverse Event | 6 | 6
Not completed — Lack of Efficacy | 2 | 6
Not completed — Loss of efficacy | 0 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Other: Loss of Patient Compliance | 0 | 1
Not completed — Other: Surgery | 0 | 1
Period: Open Label
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Started | 20 | 7
Completed | 18 | 7
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Other: Subject moved to extension study | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo | Total
Number analyzed (Participants) | 96 | 98 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 78 | 80 | 158
  >=65 years | 18 | 17 | 35
Age Continuous [Mean (Standard Deviation); unit: years] | 53.6 (11.9) | 54.0 (12.4) | 53.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 75 | 156
  Male | 15 | 23 | 38
Region of Enrollment [Number; unit: participants]
  France | 2 | 2 | 4
  Poland | 40 | 46 | 86
  Austria | 17 | 15 | 32
  Germany | 31 | 31 | 62
  Italy | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Clinical Disease Activity Index (CDAI) Remission (≤2.8) at Both Week 20 and Week 24
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in cm), and Physician's Global Assessment of Disease Activity - Visual Analog Scale (PhGADA-VAS in cm). 28 joints are examined where a lower score indicates less disease activity. Missing values were imputed using Non-Responder Imputation (NRI)
Time Frame: Week 20 and Week 24
Population: All 194 subjects in the Full Analysis Set (FAS) are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 96 | 98
percentage of subjects | 18.8 | 6.1

2. Secondary Outcome: 28-joint Count Disease Activity Score (DAS28-ESR) Remission (<2.6) at Both Week 20 and Week 24
Description: DAS28-ESR is calculated using the tender joint count (TJC), swollen joint count (SJC) erythrocyte sedimentation rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Patient Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity. Missing values were imputed using Non-Responder Imputation (NRI)
Time Frame: Week 20 and Week 24
Population: Since imputation was used, all 194 subjects are included in the analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 96 | 98
percentage of subjects | 19.8 | 3.1

3. Secondary Outcome: Simplified Disease Activity Index (SDAI) Remission (≤3.3) at Both Week 20 and Week 24
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/dL), Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in cm), and Physician's Global Assessment of Disease Activity - Visual Analog Scale (PhGADA-VAS in cm). 28 joints are examined where a lower score indicates less disease activity. Missing values were imputed using Non-Responder Imputation (NRI)
Time Frame: Week 20 and Week 24
Population: Since imputation was used, all 194 subjects are included in the analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 96 | 98
percentage of subjects | 14.6 | 4.1

4. Secondary Outcome: Time From Stopping Treatment (Week 24) to Loss of Remission (up to Week 52) Assessed Using Clinical Disease Activity Index (CDAI) Scores at 2 Consecutive Visits
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in cm), and Physician's Global Assessment of Disease Activity - Visual Analog Scale (PhGADA-VAS in cm). 28 joints are examined where a lower score indicates less disease activity. Patients losing remission (CDAI >2.8) for two consecutive visits will be considered as having the event on the day of the visit where remission was first lost. Subjects discontinued/non-remitted by Week 24 are considered as having the event on day 1.
Time Frame: Week 24 up to Week 52
Population: All 194 subjects in the Full Analysis Set (FAS) are included in this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 96 | 98
days | 12.1 (2.83) | 3.4 (1.02)

5. Secondary Outcome: Time From Stopping Treatment (Week 24) to Loss of Remission (up to Week 52) Assessed Using Simplified Disease Activity Index (SDAI) Scores at 2 Consecutive Visits
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), C-reactive protein (mg/dL), Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in cm) and Physician's Global Assessment of Disease Activity (PhGADA-VAS in cm). 28 joints are examined. A lower score indicates less disease activity. Patients losing remission (SDAI >3.3) for two consecutive visits will be considered as having the event on the day of the visit where remission was first lost. Subjects discontinued/non-remitted by Week 24 are considered as having the event on day 1.
Time Frame: Week 24 up to Week 52
Population: All 194 subjects in the Full Analysis Set (FAS) are included in this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 96 | 98
days | 9.8 (2.57) | 2.1 (0.53)

6. Secondary Outcome: Time From Stopping Treatment (Week 24) to Loss of Remission (up to Week 52) Assessed Using DAS28-ESR Scores at 2 Consecutive Visits
Description: DAS28-ESR is calculated using tender joint count (TJC), swollen joint count (SJC), erythrocyte sedimentation rate (ESR mm/hour) and Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS mm). 0.56x√(TJC) + 0.28x√(SJC) + 0.70xlognat(ESR) + 0.014xPtGADA-VAS. 28 joints are examined. Lower score indicates less disease activity. Patients losing remission (DAS28-ESR≥2.6) for two consecutive visits will be considered as having the event on the first of the two visits. Subjects discontinued/non-remitted by Week 24 are considered as having the event on day 1.
Time Frame: Week 24 up to Week 52
Population: All 194 subjects in the Full Analysis Set (FAS) are included in this analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 96 | 98
Days | 12.1 (2.96) | 1.0 (0.00)

7. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 24
Description: ACR20 responders are subjects with at least 20% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale, 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale. Missing values were imputed using Non-Responder Imputation (NRI)
Time Frame: Baseline, Week 24
Population: Since imputation was used, all 194 subjects are included in the analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 96 | 98
percentage of subjects | 36.5 | 15.3

8. Secondary Outcome: American College of Rheumatology 50% (ACR50) Response at Week 24
Description: ACR50 responders are subjects with at least 50% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale, 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale. Missing values were imputed using Non-Responder Imputation (NRI)
Time Frame: Baseline, Week 24
Population: Since imputation was used, all 194 subjects are included in the analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 96 | 98
percentage of subjects | 20.8 | 7.1

9. Secondary Outcome: American College of Rheumatology 70% (ACR70) Response at Week 24
Description: ACR70 responders are subjects with at least 70% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale, 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale. Missing values were imputed using Non-Responder Imputation (NRI)
Time Frame: Baseline, Week 24
Population: Since imputation was used, all 194 subjects are included in the analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 96 | 98
percentage of subjects | 9.4 | 3.1

10. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 24
Description: HAQ-DI is derived based on the mean of individual scores in 8 categories of daily living actives (using 20 questions). Each question is scored 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). Change from Baseline is computed as the value at Week 24 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 24
Population: Of the 194 subjects, 182 (91 CZP, 91 Placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 91 | 91
units on a scale | -0.25 (0.460) | -0.03 (0.490)

11. Secondary Outcome: Change From Baseline in Short Form 36-items Health Survey (SF-36) Physical Component Summary (PCS) Scores at Week 24
Description: PCS norm-based scores are calculated based upon the following 8 domain scores, Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health, and range from 1 to 81, where 50 represents the normative value. A larger positive value in change from Baseline indicates an improvement.
Time Frame: Baseline, Week 24
Population: Of the 194 subjects in the Full Analysis Set (FAS), 164 (82 CZP, 82 Placebo) had values at Baseline and Week 24 and are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 82 | 82
units on a scale | 6.0 (7.50) | 1.7 (7.56)

12. Secondary Outcome: Change From Baseline in Short Form 36-items Health Survey (SF-36) Mental Component Summary (MCS) Scores at Week 24
Description: MCS norm-based scores are calculated based upon the following 8 domain scores, Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health, and range from -9 to 82, where 50 represents the normative value. A larger positive value in change from Baseline indicates an improvement
Time Frame: Baseline, Week 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 82 | 82
units on a scale | 4.0 (9.77) | 0.5 (9.26)

13. Secondary Outcome: Change From Baseline in Short Form 36-items Health Survey (SF-36) Physical Functioning Domain at Week 24
Description: There are 8 SF-36 domain scores: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health, each ranging from 0 to 100, with higher scores indicating better health. A larger positive value in change from Baseline indicates an improvement
Time Frame: Baseline, Week 24
Population: Of the 194 subjects in the Full Analysis Set (FAS), 168 (83 CZP, 85 Placebo) had values at Baseline and Week 24 and are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 83 | 85
units on a scale | 5.1 (7.36) | 0.4 (8.90)

14. Secondary Outcome: Change From Baseline in Short Form 36-items Health Survey (SF-36) Role Physical Domain at Week 24
Description: as for outcome 13
Time Frame: Baseline, Week 24
Population: Of the 194 subjects in the Full Analysis Set (FAS), 167 (83 CZP, 84 Placebo) had values at Baseline and Week 24 and are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 83 | 84
units on a scale | 4.7 (9.77) | 1.7 (7.81)

15. Secondary Outcome: Change From Baseline in Short Form 36-items Health Survey (SF-36) Bodily Pain Domain at Week 24
Description: as for outcome 13
Time Frame: Baseline, Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 83 | 84
units on a scale | 8.0 (8.70) | 2.8 (8.50)

16. Secondary Outcome: Change From Baseline in Short Form 36-items Health Survey (SF-36) General Health Domain at Week 24
Description: as for outcome 13
Time Frame: Baseline, Week 24
Population: Of the 194 subjects in the Full Analysis Set (FAS), 166 (82 CZP, 84 Placebo) had values at Baseline and Week 24 and are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 82 | 84
units on a scale | 5.0 (7.59) | 0.9 (8.06)

17. Secondary Outcome: Change From Baseline in Short Form 36-items Health Survey (SF-36) Vitality Domain at Week 24
Description: as for outcome 13
Time Frame: Baseline, Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 83 | 85
units on a scale | 6.4 (8.74) | 0.6 (8.41)

18. Secondary Outcome: Change From Baseline in Short Form 36-items Health Survey (SF-36) Social Functioning Domain at Week 24
Description: as for outcome 13
Time Frame: Baseline, Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 83 | 85
units on a scale | 4.3 (10.21) | 0.8 (8.89)

19. Secondary Outcome: Change From Baseline in Short Form 36-items Health Survey (SF-36) Role Emotional Domain at Week 24
Description: as for outcome 13
Time Frame: Baseline, Week 24
Population: Of the 194 subjects in the Full Analysis Set (FAS), 166 (83 CZP, 83 Placebo) had values at Baseline and Week 24 and are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 83 | 83
units on a scale | 3.2 (13.74) | -0.2 (12.33)

20. Secondary Outcome: Change From Baseline in Short Form 36-items Health Survey (SF-36) Mental Health Domain at Week 24
Description: as for outcome 13
Time Frame: Baseline, Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 83 | 85
units on a scale | 5.2 (8.43) | 1.2 (7.72)

21. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain-Visual Analog Scale (VAS) at Week 24
Description: Change from Baseline in Patient's Assessment of Arthritis Pain-VAS (0 to 100 mm visual analog scale, 0 being no pain and 100 being most severe pain) is computed as the value at Week 24 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 24
Population: Of the 194 subjects, 162 (81 CZP, 81 Placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 81 | 81
mm | -12.4 (25.49) | 1.0 (24.27)

22. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS) at Week 24
Description: Change from Baseline in Patient's Global Assessment of Disease Activity-VAS (0 to 100 mm visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as the value at Week 24 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 24
Population: Of the 194 subjects, 183 (92 CZP, 91 Placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 92 | 91
mm | -7.6 (28.69) | 2.9 (25.43)

23. Secondary Outcome: Change From Baseline in Fatigue Assessment Scale at Week 24
Description: Change from Baseline in Fatigue Assessment scale (0 to 10, 0 is "No Fatigue" and 10 is "Fatigue as bad as you can imagine") is computed as the value at Week 24 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 24
Population: Of the 194 subjects, 180 (90 CZP, 90 Placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 90 | 90
units on a scale | -1.2 (2.24) | 0.1 (2.12)

24. Other Pre Specified Outcome: Time From Stopping Treatment (Week 24) to First Flare (up to Week 52) Using Clinical Disease Activity Index (CDAI) at 2 Consecutive Visits
Description: Subjects having a flare (CDAI ≥11) between Week 24 and Week 52 for two consecutive visits will be considered as having the event on the day of the visit where flare first appeared.
Time Frame: From Week 24 up to Week 52
Population: All 194 subjects in the Full Analysis Set (FAS) are included in this analysis.
  An ad-hoc analysis has been performed on the Week 24 Responder Set (W24RS) which showed similar results.
Measure: Mean (Standard Error); unit: days
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 96 | 98
days | 82.3 (10.28) | 34.5 (4.93)

25. Other Pre Specified Outcome: Association Between Clinical Disease Activity Index (CDAI) and Simplified Disease Activity Index (SDAI) Activity States at Week 24
Description: The number representing the association is the Kappa Correlation Coefficient for CDAI/SDAI for each category of activity (Low Disease Activity (LDA) vs. non-LDA, Medium Disease Activity (MDA) vs. non-MDA, and High Disease Activity (HDA) vs. non-HDA).
Time Frame: Week 24
Population: Of the 194 subjects in the Full Analysis Set (FAS) 143 (76 CZP, 67 Placebo) had measures for both CDAI and SDAI at Week 24 and are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Kappa Correlation Coefficient
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 76 | 67
Kappa Correlation Coefficient
  LDA vs. Non-LDA | 0.82 [0.69 to 0.95] | 0.96 [0.89 to 1.00]
  MDA vs. Non-MDA | 0.68 [0.49 to 0.87] | 0.71 [0.54 to 0.88]
  HDA vs. Non-HDA | 0.59 [0.27 to 0.90] | 0.71 [0.53 to 0.89]

26. Other Pre Specified Outcome: Association Between Clinical Disease Activity Index (CDAI) and Disease Activity Score (DAS28-ESR) Activity States at Week 24
Description: The number representing the association is the Kappa Correlation Coefficient for CDAI/DAS28-ESR for each category of activity (Low Disease Activity (LDA) vs. non-LDA, Medium Disease Activity (MDA) vs. non-MDA, and High Disease Activity (HDA) vs. non-HDA).
Time Frame: Week 24
Population: Of the 194 subjects in the Full Analysis Set (FAS) 148 (79 CZP, 69 Placebo) had measures for both CDAI and DAS28-ESR at Week 24 and are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Kappa Correlation Coefficient
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 79 | 69
Kappa Correlation Coefficient
  LDA vs. Non-LDA | 0.08 [-0.10 to 0.26] | 0.08 [-0.15 to 0.31]
  MDA vs. Non-MDA | 0.36 [0.19 to 0.54] | 0.44 [0.27 to 0.60]
  HDA vs. Non-HDA | 0.54 [0.22 to 0.85] | 0.65 [0.46 to 0.84]

27. Other Pre Specified Outcome: Association Between Disease Activity Score (DAS28-ESR) and Simplified Disease Activity Index (SDAI) Activity States at Week 24
Description: The number representing the association is the Kappa Correlation Coefficient for DAS28-ESR/SDAI for each category of activity (Low Disease Activity (LDA) vs. non-LDA, Medium Disease Activity (MDA) vs. non-MDA, and High Disease Activity (HDA) vs. non-HDA).
Time Frame: Week 24
Population: Of the 194 subjects in the Full Analysis Set (FAS) 142 (76 CZP, 66 Placebo) had measures for both DAS28-ESR and SDAI at Week 24 and are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Kappa Correlation Coefficient
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 76 | 66
Kappa Correlation Coefficient
  LDA vs. Non-LDA | 0.20 [0.03 to 0.37] | 0.10 [-0.13 to 0.33]
  MDA vs. Non-MDA | 0.44 [0.26 to 0.62] | 0.59 [0.42 to 0.77]
  HDA vs. Non-HDA | 0.74 [0.39 to 1.00] | 0.91 [0.79 to 1.00]

28. Other Pre Specified Outcome: Association Between Clinical Disease Activity Index (CDAI) and Simplified Disease Activity Index (SDAI) Remission at Week 24
Description: The number representing the association is the Kappa Correlation Coefficient for CDAI/SDAI remission.
Time Frame: Week 24
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Kappa Correlation Coefficient
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 76 | 67
Kappa Correlation Coefficient | 0.88 [0.74 to 1.00] | 1.00 [1.00 to 1.00]

29. Other Pre Specified Outcome: Association Between Clinical Disease Activity Index (CDAI) and Disease Activity Score (DAS28-ESR) Remission at Week 24
Description: The number representing the association is the Kappa Correlation Coefficient for CDAI/DAS28-ESR remission
Time Frame: Week 24
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Kappa Correlation Coefficient
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 79 | 69
Kappa Correlation Coefficient | 0.53 [0.32 to 0.75] | 0.31 [-0.07 to 0.69]

30. Other Pre Specified Outcome: Association Between Disease Activity Score (DAS28-ESR) and Simplified Disease Activity Index (SDAI) Remission at Week 24
Description: The number representing the association is the Kappa Correlation Coefficient for DAS28-ESR/SDAI remission.
Time Frame: Week 24
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Kappa Correlation Coefficient
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo
Number analyzed (Participants) | 76 | 66
Kappa Correlation Coefficient | 0.61 [0.41 to 0.81] | 0.31 [-0.08 to 0.69]

ADVERSE EVENTS:
Time Frame: The first two columns refer to the 24-week double blind (DB) phase, and an additional 12-week follow up for those not entering the open label (OL) phase. The third column displays AEs for the 28-week OL phase and a potential 12-week safety follow-up.
Description: A Treatment Emergent Adverse Event (TEAE) in the OL phase is an AE for which the onset date and time is after 84 days after last injection in the DB treatment phase and not later than the date of the last visit for non-retreated patients or not later than 84 days after last injection for retreated patients.
Groups:
- Open Label Phase: At Week 24 subjects are evaluated. Non-remitters are discontinued from the study with the opportunity to enter another open label (OL) study. Remitters stop randomized treatment and are followed up until Week 52. Remitters who flare up between Week 24 and Week 52 will be re-treated with (3 administrations of 400 mg CZP, given every other week, followed by 200 mg CZP given every other week) up to and including Week 50. Of the 27 subjects in the OL phase 15 were retreated and 12 were not retreated.
Arm/Group | Certolizumab Pegol 200 mg (CDP870) | Placebo | Open Label Phase
Serious Adverse Events (participants affected / at risk) | 5/96 | 7/98 | 1/27
Other Adverse Events (participants affected / at risk) | 32/96 | 34/98 | 4/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol 200 mg (CDP870) (N=96) | Placebo (N=98) | Open Label Phase (N=27)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haemophilus Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) — The Cerebrovascular Accident occurring during the open label (OL) phase occurred in a subject who did not receive treatment throughout the duration of the OL phase.
Wegener's Granulomatosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol 200 mg (CDP870) (N=96) | Placebo (N=98) | Open Label Phase (N=27)
Nasopharyngitis (Infections and infestations) | 10 (12) | 11 (13) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (6) | 4 (5) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 6 (6) | 5 (5) | 0 (0)
Bronchitis (Infections and infestations) | 3 (4) | 5 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 6 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (6) | 2 (2)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 5 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.